CLINICAL TRIAL: NCT05148520
Title: Provision of Service of a Youth Quitline Programme For Youth Smokers
Brief Title: Provision of Service of a YQL Programme For Youth Smokers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: YQL
Record Dates: First submitted 2021-11-25; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Mental Health Issue
Keywords: smoking cessation service; youth smoker

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 5A's model (Other): The practice guideline emphasizes on the use of '5A's' model that contains five major steps in providing smoking cessation counselling. Specifically, our counsellors will take the following steps to provide telephone counselling for youth smokers who are ready to quit smoking
  Interventions: Behavioral: 5A's model

INTERVENTIONS:
Behavioral: 5A's model — (1) Ask - ask youth smokers about their smoking habit, (2) Advise - advise youth smokers to quit smoking, (3) Assess - assess youth smokers about their willingness to quit smoking, (4) Assist - assist youth smokers who are willing to make a quit attempt, and (5) Arrange
  - arrange for follow-up.

SUMMARY:
This project is funded by Department of Health. We will run a quitline which provides telephone smoking cessation counseling to youth smokers aged 25 or below. After baseline counseling based on trans-theoretical model, follow-up counseling will be provided by trained counselors (i.e. nursing students or students from other healthrelated disciplines) at 1 week, 1, 3, 6, 9 and 12 months. It is expected that the quitline can assist youth smokers to quit smoking, thus saving the healthcare cost attributed to smoking in long-term.

DETAILED DESCRIPTION:
This project will last for 15 months (from 1st Dec 2020 to 28th Feb 2022). Prior to commencement, a month will be spent on preparation, including setting up the quitline and website, designing and printing publicity materials, connecting with secondary and post-secondary schools and training peer counsellors. We will operate the quitline for 15 months and provide telephone counselling for eligible youth smokers. Self-reported quitters at 6-month follow-up will be invited for biochemical validation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 or below
* Self-reported to smoke any types of tobacco products within the past 1 month
* Speak Cantonese and
* Provide verbal consent to counselling service.

Exclusion Criteria:

* have psychiatric disease
* and/or currently receive any smoking cessation intervention from other service providers

Max Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Self-reported 7-point prevalence | at the 6-month follow-up
  The self-reported abstinence will be validated if the level of carbon monoxide in expired air was less than 4 parts per million and saliva cotinine level was less than100 ng/mL in parallel tests.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yan Ho, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Ka Yan Ho, Hong Kong, Hong Kong,China, Hong Kong